CLINICAL TRIAL: NCT04000789
Title: The Effect of Combination of Vitamin A, Vitamin E, Sodium Hyaluronate 0.15% Eye Drop Compared With Sodium Hyaluronate 0.1% Eye Drop to Tear Film Stability and Conjunctival Goblet Cells Density in Patient With Non-Proliferative Diabetic Retinopathy (NPDR), and Proliferative Diabetic Retinopathy (PDR)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dr Cipto Mangunkusumo General Hospital (Other)
Responsible Party: Principal Investigator, Made Susiyanti, dr., Dr Cipto Mangunkusumo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19-06-0740
Record Dates: First submitted 2019-06-26; First posted 2019-06-27 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Non-Proliferative Diabetic Retinopathy; Proliferative Diabetic Retinopathy New Vessels on Disc; Dry Eye Syndromes
Keywords: Diabetes Mellitus; Proliferative Diabetic Retinopathy; Non-Proliferative Diabetic Retinopathy; Dry Eye Syndromes; Sodium Hyaluronate; Vitamin A; Vitamin E
MeSH Terms: conditions — Dry Eye Syndromes; Diabetes Mellitus | interventions — Hyaluronic Acid; Vitamin A; Vitamin E

STUDY DESIGN:
Intervention Model Description: The study examining DM patient with NPDR or PDR complication with decrease corneal sensitivity. Patient with decreased corneal sensitivity were grouped between NPDR and PDR. NPDR group divided into treatment group (combination of sodium hyaluronate, vitamin A and Vitamin E eye drops given 6 times/day) and control group (Sodium Hyaluronate eye drops only given 6 times/day). Likewise, PDR group divided into treatment group (combination of sodium hyaluronate, vitamin A and Vitamin E eye drops given 6 times/day) and control group (Sodium Hyaluronate eye drops only given 6 times/day).
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- NPDR (Experimental)
  Interventions: Drug: Sodium Hyaluronate, Vitamin A, Vitamin E
- NPDR Comparator (Active Comparator)
  Interventions: Drug: Sodium Hyaluronate, Vitamin A, Vitamin E
- PDR (Experimental)
  Interventions: Drug: Sodium Hyaluronate, Vitamin A, Vitamin E
- PDR Comparator (Active Comparator)
  Interventions: Drug: Sodium Hyaluronate, Vitamin A, Vitamin E

INTERVENTIONS:
Drug: Sodium Hyaluronate, Vitamin A, Vitamin E — Eye drops consisting of combination of Sodium Hyaluronate, Vitamin A, Vitamin E will be . given to patients in control groups

SUMMARY:
Commonly know that one of the complications caused by Diabetes Mellitus (DM) is microangiopathy. Microangiopathy in the long term may lead to neuropathy of the corneal nerves. Neuropathy of the cornea will lead to dry eyes in DM patient. One of the artificial tears used in treating dry eyes is sodium hyaluronate. But until recently no research had been done in examining the effect of giving combination of sodium hyaluronate, vitamin A and vitamin E in dry eyes. The antioxidant, and capability of vitamin A and E in promoting cell proliferation may alleviate the symptoms of dry eyes. In this paper we used Ocular Surface Disease Index (OSDI), Tear Break Up time, Schirmer I test and impression cytology to assess baseline and 28 days post therapy in patient with Non-Proliferative Diabetic Retinopathy (NPDR), and Proliferative Diabetic Retinopathy (PDR)

DETAILED DESCRIPTION:
The study is double blind randomized clinical trial, comparing the usage of combination of sodium hyaluronate 0.15%, vitamin A and vitamin E eye drops compared to sodium hyaluronate 0.1% eye drop only in patient with NPDR or PDR with decreased corneal sensitivity. The examination consisted of OSDI questionnaire, tear film break up time, Schirmer I, and goblet cell density, examined at baseline and 4 weeks (day 28) after the initial eye drops is given. For sample size calculation, estimated 96 patients are required to give statistical effect, this number already calculating the possibility of 20% drop out rate. Every eligible patient is then randomized with block randomization into each allocated arm. Statistical analysis used for this study is unpaired T test if the data distribution is normal, if not Mann-Whitney test will be used.

ELIGIBILITY:
Inclusion Criteria:

* DM patients with NPDR or PDR
* Corneal sensitivity less than 45 mm with Cochet Bonnet esthesiometer

Exclusion Criteria:

* Patient with anterior chamber inflammation
* Patient with history of ocular surgery (ex. Repair of corneal rupture, cataract surgery, Lasik)
* Patient with history of cerebrovascular event that may affect cognitive function
* Patient had event of disease which may impact corneal sensitivity (ex. Viral keratitis, ophthalmic Herpes Zoster)
* Patient with corneal cicatrix
* Patient on anti-allergic medication
* Pregnant or lactating woman

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2019-07 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Ocular Surface Disease Index (OSDI) questionnaire | 4 weeks
  A questionnaire to measure subjective symptoms of dry eyes. Possible score of 0 (no dry eye) to 100 (severe dry eye). Measured at baseline, day 14 and day 28.
Tear Film Breakup Time | 4 weeks
  Measurement in seconds of tear film stability. The shorter the fluorescein tear break up time, the lower the tear film stability. Measured at baseline and day 28.
Schirmer I Test | 4 weeks
  Measurement of tear production. The amount of tears are measured in total millimeters after 5 minutes has elapsed. Measured at baseline and day 28.
Conjunctival Goblet Cell Density | 4 weeks
  Measurement of conjunctival goblet cell count per mm2. Measured at baseline and day 28.

IPD SHARING:
Plan to Share IPD: No